CLINICAL TRIAL: NCT00445822
Title: Protocol for Standardized Diagnostic Procedures, Registration, and Treatment Recommendations in Children and Adolescents With Philadelphia Chromosome-positive Chronic Myeloid Leukemia (CML)
Brief Title: Registration of Children With CML and Treatment With Imatinib
Acronym: CML-paed II
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Technische Universität Dresden (Other)
Collaborators: Medical Academy of Wroclaw, Poland (Unknown); University of Leiden, Netherlands (Unknown); Nordic Society for Pediatric Hematology and Oncology (Other); University of Genua, Italy (Other)
Responsible Party: Prof. Dr. Meinolf Suttorp, Universitätskinderklinik Dresden
Other Study IDs: TUD-CML-paed 016; EudraCT: 2007-001339-69
Record Dates: First submitted 2007-03-08; First posted 2007-03-09 (Estimated); Last update posted 2012-02-29 (Estimated); Status verified 2012-02

CONDITIONS: Myeloid Leukemia, Chronic
Keywords: CML; Children; Imatinib; bcr-abl; Response; Imatinib mesylate
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Bone Marrow and blood smears
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Newly diagnosed pediatric patients (age < 19 years) with bcr-abl-positive CML will be treated with imatinib. Serial monitoring of treatment response is performed in one month intervals during the first three months of treatment and in three months intervals thereafter. Patients with non-response, poor response (either molecular, cytogenetic, or hematologic non-/poor response) or progress of the disease while under imatinib treatment will stop imatinib and undergo stem cell transplantation. All responders to imatinib treatment with an HLA matched donor will undergo stem cell transplantation not later than 2 years after diagnosis.

DETAILED DESCRIPTION:
Indication:

Newly diagnosed pediatric patients with bcr-abl-positive CML.

Design:

Multicenter, non-randomized, open, prospective clinical trial.

Objectives:

Primary:

- assessment of antileukemic activity of imatinib in children and adolescents with Philadelphia chromosome-positive chronic myeloid leukemia

Secondary:

* assessment of the time-to event-efficacy variables
* correlation of the quality of haematological, cytogenetical and molecular remission in children and adolescents with CML on ongoing imatinib therapy with survival
* safety of imatinib

Endpoints:

Primary:

- rate of haematological, cytogenetical and molecular remissions

Secondary:

* time to progression
* duration of chronic phase
* time to loss of response
* overall survival
* assessment of treatment-related toxicities in children and adolescents.

Inclusion criteria:

Newly diagnosed Ph+ or bcr-abl-positive CML- Male and female patients aged 0 to 18 years- Written informed consent

Exclusion criteria:

* CML without bcr-abl rearrangement detectable by PCR
* Pretreatment with Interferon alpha or any other cytostatic drug with the exception of hydroxyurea or anagrelide (Note: anagrelide is not approved in Germany for treatment of CML). However, these patients may be registered as observational patients.
* Any other severe underlying disease beside CML.
* Age > 18 years
* Pregnant or lactating women
* Subjects unlikely to comply with the requirements of the protocol

Number of patients to be enrolled: 150

Recruitment period: 5 years

Treatment period: 2 years

Planned start of study: 2007

Planned end of study: 2013

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed Ph+ or bcr-abl-positive CML
* Male and female patients aged 0 to 18 years
* Written informed consent

Exclusion Criteria:

* CML without bcr-abl rearrangement detectable by PCR
* Pretreatment with Interferon alpha or any other cytostatic drug with the exception of hydroxyurea or anagrelide (Note: anagrelide is not approved in Germany for treatment of CML). However, these patients may be registered as observational patients.
* Any other severe underlying disease beside CML.
* Age > 18 years- Pregnant or lactating women
* Subjects unlikely to comply with the requirements of the protocol

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pts younger than 19 years with PH+ CML are recruited from primary care clinics
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2007-03; Primary Completion 2012-07 (Estimated); Study Completion 2012-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Meinolf Suttorp, Prof. Dr., Principal Investigator — University Children's Hospital, Dpt. Ped. Hemato-Oncology, Technical University of Dresden, Germany
Locations (1):
- University Children's Hopsital, Technical University of Dresden, Fetscherstr. 74, Dresden, Saxony, Germany

REFERENCES:
- [Background] Millot F, Guilhot J, Nelken B, Leblanc T, De Bont ES, Bekassy AN, Gadner H, Sufliarska S, Stary J, Gschaidmeier H, Guilhot F, Suttorp M. Imatinib mesylate is effective in children with chronic myelogenous leukemia in late chronic and advanced phase and in relapse after stem cell transplantation. Leukemia. 2006 Feb;20(2):187-92. doi: 10.1038/sj.leu.2404051. PMID 16341042
- [Background] Adler R, Viehmann S, Kuhlisch E, Martiniak Y, Rottgers S, Harbott J, Suttorp M. Correlation of BCR/ABL transcript variants with patients' characteristics in childhood chronic myeloid leukaemia. Eur J Haematol. 2009 Feb;82(2):112-8. doi: 10.1111/j.1600-0609.2008.01170.x. Epub 2008 Nov 10. PMID 19067742
- [Background] Suttorp M. Innovative approaches of targeted therapy for CML of childhood in combination with paediatric haematopoietic SCT. Bone Marrow Transplant. 2008 Oct;42 Suppl 2:S40-6. doi: 10.1038/bmt.2008.282. PMID 18978743
- [Background] Schmid H, Jaeger BA, Lohse J, Suttorp M. Longitudinal growth retardation in a prepuberal girl with chronic myeloid leukemia on long-term treatment with imatinib. Haematologica. 2009 Aug;94(8):1177-9. doi: 10.3324/haematol.2009.008359. Epub 2009 Jun 22. No abstract available. PMID 19546438
- [Background] Bacher U, Klyuchnikov E, Zabelina T, Ottinger H, Beelen DW, Schrezenmeier H, Ehninger G, Muller C, Berger J, Suttorp M, Kolb HJ, Kroger N, Zander AR. The changing scene of allogeneic stem cell transplantation for chronic myeloid leukemia--a report from the German Registry covering the period from 1998 to 2004. Ann Hematol. 2009 Dec;88(12):1237-47. doi: 10.1007/s00277-009-0737-3. Epub 2009 Mar 25. PMID 19319532
- [Background] Suttorp M, Millot F. Treatment of pediatric chronic myeloid leukemia in the year 2010: use of tyrosine kinase inhibitors and stem-cell transplantation. Hematology Am Soc Hematol Educ Program. 2010;2010:368-76. doi: 10.1182/asheducation-2010.1.368. PMID 21239821
- [Background] Suttorp M, Yaniv I, Schultz KR. Controversies in the treatment of CML in children and adolescents: TKIs versus BMT? Biol Blood Marrow Transplant. 2011 Jan;17(1 Suppl):S115-22. doi: 10.1016/j.bbmt.2010.09.003. PMID 21195300
- [Background] Suttorp M, Claviez A, Bader P, Peters C, Gadner H, Ebell W, Dilloo D, Kremens B, Kabisch H, Fuhrer M, Zintl F, Gobel U, Klingebiel T. Allogeneic stem cell transplantation for pediatric and adolescent patients with CML: results from the prospective trial CML-paed I. Klin Padiatr. 2009 Nov-Dec;221(6):351-7. doi: 10.1055/s-0029-1239529. Epub 2009 Nov 4. PMID 19890786
- [Background] Suttorp M, Tauer JT, Millot F: Chronic myeloid leukemia in children: diagnostics and management Onkologie (CZ) 5(2):12-15, 2011
- [Result] Suttorp M, Thiede C, Tauer JT, Range U, Schlegelberger B, von Neuhoff N. Impact of the type of the BCR-ABL fusion transcript on the molecular response in pediatric patients with chronic myeloid leukemia. Haematologica. 2010 May;95(5):852-3. doi: 10.3324/haematol.2009.019224. Epub 2010 Feb 9. No abstract available. PMID 20145269
- [Derived] Stiehler S, Sembill S, Schleicher O, Marx M, Rauh M, Krumbholz M, Karow A, Suttorp M, Woelfle J, Maj C, Metzler M. Imatinib treatment and longitudinal growth in pediatric patients with chronic myeloid leukemia: influence of demographic, pharmacological, and genetic factors in the German CML-PAED cohort. Haematologica. 2024 Aug 1;109(8):2555-2563. doi: 10.3324/haematol.2023.284668. PMID 38497150
- [Derived] Knofler R, Lange BS, Paul F, Tiebel O, Suttorp M. Bleeding signs due to acquired von Willebrand syndrome at diagnosis of chronic myeloid leukaemia in children. Br J Haematol. 2020 Mar;188(5):701-706. doi: 10.1111/bjh.16241. Epub 2019 Oct 15. PMID 31617211
- [Derived] Ulmer A, Tabea Tauer J, Glauche I, Jung R, Suttorp M. TK inhibitor treatment disrupts growth hormone axis: clinical observations in children with CML and experimental data from a juvenile animal model. Klin Padiatr. 2013 May;225(3):120-6. doi: 10.1055/s-0033-1343483. Epub 2013 May 28. PMID 23716272
- [Derived] Jaeger BA, Tauer JT, Ulmer A, Kuhlisch E, Roth HJ, Suttorp M. Changes in bone metabolic parameters in children with chronic myeloid leukemia on imatinib treatment. Med Sci Monit. 2012 Dec;18(12):CR721-8. doi: 10.12659/msm.883599. PMID 23197234